CLINICAL TRIAL: NCT00882401
Title: The Effect of Vitamin D on the Microcirculation of Patients With Chronic Kidney Disease (CKD) and Vitamin D Deficiency
Brief Title: Vitamin D, Chronic Kidney Disease (CKD) and the Microcirculation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Dr Gavin Dreyer, Barts & The London NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-008745-38; EUDRACT number 2008-008745-38
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Kidney Disease; Vitamin D Deficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vitamin D Deficiency | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergocalciferol (oral) (Active Comparator): ergocalciferol: 50,000 IU per week for 1 month followed by 50,000 IU per month for 5 months.
  Interventions: Drug: Ergocalciferol (Vitamin D)
- Placebo (Placebo Comparator): Matching placebo at same dose schedule as ergocalciferol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergocalciferol (Vitamin D) — ergocalciferol: 50,000 IU per week for 1 month followed by 50,000 IU per month for 5 months.
  Other Names: Drisdol
  Arms: Ergocalciferol (oral)
Drug: Placebo — Matching placebo at same dose schedule as ergocalciferol
  Arms: Placebo

SUMMARY:
Overall research aims: This study will examine the effect of vitamin D supplementation on the function of the endothelium and microcirculation of patients with chronic kidney disease and vitamin D deficiency.

Hypothesis: Vitamin D therapy in patients with CKD and concomitant vitamin D deficiency will improve endothelial, and therefore microcirculatory function, reduce levels of oxidative stress and thus reduce the risk of future CVS events in this population.

DETAILED DESCRIPTION:
Research rationale: Cardiovascular (CVS) diseases are the major cause of death in patients with chronic kidney disease (CKD), accounting for approximately half of all deaths. Patients with CKD are far more likely to die of CVS disease than progress to end stage renal disease. Recently, vitamin D deficiency has been identified as a non-traditional CVS risk factor. However, vitamin D is not routinely prescribed in the early stages of CKD.

Previous publications have established that endothelial, and therefore, microcirculatory dysfunction is a marker of CVS health and a predictor of future CVS events. Studies have also shown that clinical assessments of the microcirculation reflect the overall health and function of the endothelium. Vitamin D has been shown to improve endothelial function in diabetic patients with vitamin D deficiency and normal kidney function. However, no study has examined endothelial dysfunction in patients with CKD and vitamin D deficiency.

With the prevalence of CKD and concomitant vitamin D deficiency increasing worldwide, there is a pressing need to examine the effects of vitamin D therapy in the early stages of CKD. This study involves the use of four, non-invasive, detailed assessments of the microcirculation which could be used in a clinical setting to enhance CVS risk profiling. The current study design includes novel clinical and in vitro work examining endothelial function, oxidative stress levels and potential cellular mechanisms by which vitamin D improves endothelial function. Early detection of endothelial dysfunction, before end stage renal disease is reached, will provide a powerful tool for predicting future CVS events and thus provide an opportunity to intervene with therapies, including vitamin D, at an early stage of renal dysfunction.

Study objectives: Primary study objective - to evaluate the effects of vitamin D therapy on endothelial function in patients with CKD and vitamin D deficiency. Secondary study objective: to evaluate the effects of vitamin D therapy on key clinical parameters in patients with CKD and vitamin D deficiency.

Research plan: We will conduct a double blind, randomised control trial comparing oral ergocalciferol to a placebo in adult, non-diabetic patients with CKD stages 3-4 and vitamin D deficiency (defined as < 10ng/ml (<30nmol/L)). Based on power calculations, 40 subjects will be recruited in each arm as well as 15 healthy control subjects. Subjects will be followed for 7 months in total.

ELIGIBILITY:
Inclusion Criteria:

1. eGFR between 15 and 60 ml/min/1.73m2
2. Serum 25 (OH) vitamin D levels <30nmol/L
3. No evidence of diabetes mellitus (fasting blood sugar <7.1, not taking any diabetic medication)
4. Not receiving haemo or peritoneal dialysis
5. No dialysis therapy within the last 3 months
6. Age > 18 years and < 80 years
7. Patient agrees not use any medications (prescribed or over-the-counter including herbal remedies) judged to be clinically significant by the Principal Investigator during the course of the study.
8. Able to understand and sign the written Informed Consent Form.
9. Able and willing to follow the Protocol requirements.

Exclusion Criteria:

1. Currently receiving oral ergocalciferol at any dose
2. Received IM ergocalciferol therapy within last 3 months
3. Receiving renal replacement therapy of any type or having recently received any form of dialysis (within 3 months)
4. Pacemaker or any other implanted cardiac device
5. Serum calcium above 2.6 mmol/L at screening
6. Pregnant or lactating
7. Known hypersensitivity to ergocalciferol
8. Patient known to have a condition which predisposes to hypercalcaemia (multiple myeloma, sarcoidosis, other granulomatous disease)
9. Initial blood pressure of >160/100 mmHg
10. History of significant liver disease or cirrhosis
11. Anticipated requirement for dialysis in 6 months
12. Malabsorption, severe chronic diarrhea, or ileostomy
13. Known diagnosis of hypervitaminosis D
14. Known to have diabetes mellitus
15. Known to have renal calculi
16. Known to have systemic sclerosis, Raynaud's phenomenon or other disease associated with known microcirculatory dysfunction
17. Concurrent participation in any other research study
18. Unwilling or unable to complete study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Microcirculatory function - iontophoresis | 6 months

SECONDARY OUTCOMES:
Key clinical parameters of CKD management | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Magdi Yaqoob, MB ChB, Study Chair — Barts and the London NHS Trust
Locations (1):
- Barts and the London NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Dreyer G, Tucker AT, Harwood SM, Pearse RM, Raftery MJ, Yaqoob MM. Ergocalciferol and microcirculatory function in chronic kidney disease and concomitant vitamin d deficiency: an exploratory, double blind, randomised controlled trial. PLoS One. 2014 Jul 9;9(7):e99461. doi: 10.1371/journal.pone.0099461. eCollection 2014. PMID 25006678